CLINICAL TRIAL: NCT00976664
Title: Orthotic Use for Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Health Sciences (Other)
Collaborators: Foot Levelers, Inc. (Industry)
Responsible Party: Principal Investigator, Jerrilyn Cambron, DC, PhD, Research and Professor in Dept of Research, National University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NUHS IRB H-0904
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Results first posted 2014-11-17 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-03

CONDITIONS: Chronic Low Back Pain
MeSH Terms: interventions — Foot Orthoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Orthotic group (Active Comparator): Subjects are asked to wear custom-made shoe orthotics for a 12 week study period.
  Interventions: Device: Shoe orthotic
- Shoe Orthotic Wait group (Other): The group serves as a cross-over control group. Subjects are asked to avoid any new therapies for the first 6 weeks of the 12 week study and during the last 6 weeks they are fitted for the custom-made shoe orthotics.
  Interventions: Device: Shoe Orthotic Wait Group

INTERVENTIONS:
Device: Shoe orthotic — Shoe orthotics are devices worn in the shoe to modify the patient's stance and gait.
  Arms: Orthotic group
Device: Shoe Orthotic Wait Group — This group receives the custom-made shoe orthotics at week 6 of the 12 week treatment program rather than week 1.
  Arms: Shoe Orthotic Wait group

SUMMARY:
The purpose of this research study is to determine the change in perceived levels of pain and dysfunction in 50 patients with chronic low back pain, following the use of custom-made shoe orthotics for a three month period. The hypothesis of this study is that custom orthotic intervention will improve the patients' low back pain and dysfunction symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females must be at least 18 years old.
2. Subjects must be symptomatic with current pain between T12 and the Sacroiliac joints with or without radiating pain.
3. Symptoms must have been present for at least three months.

Exclusion Criteria:

1. Use of custom-made shoe orthotics in the past year
2. Brain disorders (i.e.: dementia or Alzheimer's Disease) that would lead to difficulty in questionnaire completion.
3. Active conservative care (such as physical therapy or chiropractic care) for the low back received in the last six months (excluding the use of oral medications or daily at-home exercises for general well-being). We do not want to over-treat the patient or have any cross-over effects within this study from previous treatment.
4. Not fluent or literate in the English language. We will not be able to provide multiple translators within this pilot study.
5. Current or future litigation for low back pain.
6. Chronic pain other then low back pain such as fibromyalgia
7. Low back surgery in last six months.
8. Other conditions that may affect the outcomes of this study or exclude patients from participation in the study, including contraindications to orthotic use.
9. Peripheral neuropathy due to disorders such as diabetes.
10. Low back or leg pain that is not reproducible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-06; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerrilyn Cambron, DC, MPH, PhD, Principal Investigator — National University of Health Sciences
Locations (1):
- National University of Health Sciences, Lombard, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited 50 patients with chronic low back pain through media advertising in a midwestern suburban area.
Pre-assignment Details: 143 people were screened by phone, eligible patients (58) attended a baseline visit. Subjects were eligible if they were 18+ years of age and symptomatic with pain between T12-S1 joints with or without radiating pain for at least 3 months. Patients were randomized to a treatment group receiving custom-made orthotics or a wait-list control group.
Groups:
- Orthotic Group: This group received orthotics at randomization visit. Various outcome measures were collected over 12 weeks.
- Wait Group: This group received NO orthotics at the randomization group, as they were randomized to the wait-control group. Orthotics were given to these subjects at week 6. Various outcome measures were collected during the 12 weeks.
Period: Overall Study
Arm/Group | Orthotic Group | Wait Group
Started | 25 | 25
Completed | 22 | 24
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Orthotic Group | Wait Group | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Customized [Mean (Standard Deviation); unit: years]
  Age, Customized | 51 (16) | 53 (16) | 52 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 10 | 12 | 22
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS)
Description: This scale measures pain on a scale of 0 (no pain) to 10 (worst pain imaginable). A higher score on this scale indicates a worse outcome or increase in pain.
Time Frame: Randomization, Week 6, and Week 12
Population: Three participants were lost to follow-up in the Orthotic group and one was lost to follow-up in the Wait group, resulting in a drop from 25 participants in each group to 22 and 24 respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Orthotic Group | Wait Group
Number analyzed (Participants) | 22 | 24
units on a scale
  Randomization | 5.0 (2.2) | 4.3 (1.9)
  Week 6 | 2.8 (2.6) | 4.1 (2.3)
  Week 12 | 2.7 (2.5) | 2.9 (2.3)
Statistical Analysis 1: Comparison: Orthotic Group vs Wait Group; Test type: Superiority or Other; p = .0007, Wilcoxon (Mann-Whitney); Group differences in VAS for low back pain from randomization visit to 6-week visit were assessed via the Wilcoxon rank sums test
Statistical Analysis 2: Comparison: Orthotic Group vs Wait Group; Test type: Superiority or Other; p = .3913, Wilcoxon (Mann-Whitney); Group differences in VAS for low back pain from randomization visit to 12-week visit were assessed via the Wilcoxon rank sums test

2. Primary Outcome: Oswestry Disability Index (ODI)
Description: This index measures the functional disability of the subject, points on this index can range from 0-50. A higher numeric value on this scale indicates a worse outcome or increased disability (e.g. 0-10: minimal disability; 11-20: moderate disability; 21-30: severe disability; 31-50: crippling). Absolute scores are reported in the data table.
Time Frame: Randomization, Week 6, and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Orthotic Group | Wait Group
Number analyzed (Participants) | 22 | 24
units on a scale
  Randomization | 10.0 (4.9) | 10.4 (5.8)
  Week 6 | 6.2 (5.2) | 10.2 (5.4)
  Week 12 | 6.1 (5.3) | 8.9 (5.5)
Statistical Analysis 1: Comparison: Orthotic Group vs Wait Group; Test type: Superiority or Other; p = .002, Wilcoxon (Mann-Whitney); Group differences in ODI for low back pain from randomization visit to 6-week visit were assessed using the Wilcoxon rank sums test
Statistical Analysis 2: Comparison: Orthotic Group vs Wait Group; Test type: Superiority or Other; p = .0336, Wilcoxon (Mann-Whitney); Group differences in ODI for low back pain from randomization visit to 12-week visit were assessed using the Wilcoxon rank sums test

ADVERSE EVENTS:
Arm/Group | Orthotic Group | Wait Group
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

LIMITATIONS AND CAVEATS:
Subjects and clinicians were not blind to group. Subjects came from 1 region of the US, majority were white and ~50 years old. One type of orthotic was used as the only form of care. Several subjects felt discomfort/stiffness rather than pain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No